CLINICAL TRIAL: NCT04307602
Title: Long-term Exercise Effects from Robotic Walking Among Children with Severe Cerebral Palsy
Brief Title: Long-term Exercise Effects from Robotic Walking
Acronym: LEER
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Lund University (Other)
Collaborators: The Swedish Research Council (Other Government); Region Skane (Other); Halmstad University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: LU2019LEER; 2018-02433 (Other Grant/Funding Number: Swedish Research Counsil); 2019-00106 (Other: Ethical review agency); 2022-00729 (Other Grant/Funding Number: Swedish Research Counsil)
Record Dates: First submitted 2020-03-09; First posted 2020-03-13 (Actual); Last update posted 2024-09-25 (Actual); Status verified 2024-09

CONDITIONS: Exercise; Children; Cerebral Palsy
Keywords: Physical Activity; Physical Fitness; Physical Exertion; Health
MeSH Terms: conditions — Motor Activity; Cerebral Palsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Children with cerebral palsy GMFCS IV-V (Experimental): Exercise intervention in the waling aide Innowalk
  Interventions: Other: Exercise - High Intensity Interval Training (HIIT); Other: Exercise - Submaximal Steady State Training (SST)
- Children with cerebral palsy GMFCS I-II (Active Comparator): Exercise intervention on spinning bikes
  Interventions: Other: Exercise - High Intensity Interval Training (HIIT); Other: Exercise - Submaximal Steady State Training (SST)
- Children without disabilities (Active Comparator): Exercise intervention on spinning bikes
  Interventions: Other: Exercise - High Intensity Interval Training (HIIT); Other: Exercise - Submaximal Steady State Training (SST)

INTERVENTIONS:
Other: Exercise - High Intensity Interval Training (HIIT) — Exercise in the walk aid Innowalk for children for children with CP GMFCS IV-V, Exercise on spinning bike for children with CP GMFCS I-II and non-disabled children
Other: Exercise - Submaximal Steady State Training (SST) — Exercise in the walk aid Innowalk for children for children with CP GMFCS IV-V, Exercise on spinning bike for children with CP GMFCS I-II and non-disabled

SUMMARY:
The vision of the Long-term Exercise Effects from Robotic Walking (LEER) research program is to develop optimal, individualized exercise strategies that would in turn enhance the health and well-being of non-ambulatory children with cerebral palsy (CP).

To date, it has not been possible to study exercise among non-ambulatory children with cerebral palsy in a structured and standardized manner. Improved possibilities to carry out such studies are now offered by the robotic medical device Innowalk, which allows various training options in an upright weight-bearing position. In order to design optimal exercise strategies for children with cerebral palsy, the investigators will examine the effects of two tailored training programs, using Innowalk. Changes in cardiopulmonary and metabolic parameters, and in the levels of brain derived neurotropic factor (BDNF), nerve growth factor (NGF) and vascular endothelial growth factor (VEGF) will be examined.

The investigators will assess the acute (1 day), adaptive (16 weeks), and long-term (1 year) effects of the exercise programs through indirect calorimetry and blood samples at multiple time points. The investigators will also study the environmental and behavioral factors facilitating and hindering participation in exercise, by semi-structured interviews.

The goal is to design improved individualized exercise programs that will increase health and well-being in the children and their families, thereby decreasing the use of medications and healthcare.

DETAILED DESCRIPTION:
A randomized controlled intervention trial with a crossover design with a one-year follow-up will be performed to explore the differential acute and long-term effects of A) high intensity interval training (HIIT) and of B) steady state training (SST) among non-ambulatory children with CP, ambulatory children with CP and non-disabled children. Non-ambulatory children with CP will walk in the robotic medical device Innowalk. Ambulatory children with CP and non-disabled children will cycle on a cycle ergometer. As the numbers of eligible children in Skåne County, Sweden, are low and due to heterogeneity among the children with CP, a crossover design is chosen to maximize statistical power.

Aim 1: Acute response to exercise Objectives: The aim is to elucidate the acute effects form one bout of SST and one bout of HIIT in the three groups of children.

Research question: Are there differences in the physiological responses in BDNF, NGF, VEGF and metabolic bio-markers from one acute bout of HIIT and one acute bout of SST exercise among non-ambulatory children with CP, ambulatory children with CP and non-disabled children? Methodology: Indirect calorimetry will be used during one acute bout of HIIT exercise and SST exercise to assess markers of ventilation, circulation, fat versus carbohydrate oxidation, and energy expenditure during exercise. Blood will be collected before and after the exercise testing to assess differences in BDNF, NGF, VEGF and metabolic bio-markers. Temperature at the feet will be assessed to analyze vasodilation.

Deliverables: To demonstrate biomarkers of cardiopulmonary and metabolic function and BDNF, NGF, VEGF, that are the most effected by one bout of HIIT and one bout of SST among non-ambulatory children with CP, ambulatory children with CP and non-disabled children and to elucidate if there are differences between the three groups of children.

Aim 2: Adaptation to exercise Objectives: The aim is to elucidate the adaptation to 16 weeks of two types of structured training regimes (HIIT vs. SST) on cardiopulmonary and metabolic parameters and BDNF, NGF, VEGF, in the three groups of children.

Research question: Are there differences in the physiological adaptation to HIIT exercise and SST exercise among non-ambulatory children with CP, ambulatory children with CP and non-disabled children? Methodology: We will use supervised exercise training of 16 weeks with HIIT -16 weeks Washout -16 weeks with SST, starting and ending with the exercise testing described in Aim 1 to evaluate adaptation to HIIT and SST.

Deliverables: To demonstrate changes in cardiopulmonary and metabolic parameters and BDNF, NGF, VEGF in adaptation to HIIT and SST and to elucidate whether there are differences between HIIT and SST among the three groups of children.

Aim 3: Adherence to physical activity and exercise; child-family perspective Objectives: The aim is to study the adherence to the two exercise regimes among non-ambulatory children with CP, ambulatory children with CP and non-disabled children and to elucidate health and well-being factors for the child and their family.

Research question: Which are the facilitating and hindering factors to participate in structured and standardized exercise regimes and which factors are affecting health and well-being within a child-family perspective, professional caregivers and the child-family perspective and the within the healthcare system? Methodology: The methods used will be a combination of questionnaires and semi-structured interviews individually and in focus groups.

Deliverables: Description of facilitating and hindering factors for adherence in the exercise regimes among the three groups of children, and furthermore a description of factors facilitating and hindering health and well-being.

Aim 4: Long-term effects from exercise Objectives: The aim is to study the physiological long-term effects of the exercise intervention programs at a one-year follow-up and the adherence to exercise among non-ambulatory children with CP, ambulatory children with CP and non-disabled children.

Research question: Which are the physiological adaptations to exercise and which are the facilitating and hindering factors to long-term participation in exercise regimes? Methodology: The methods in Aim 1 and Aim 3 will be used to answer the research question.

Deliverables: Description of long-term physiological effects from exercise and facilitating and hindering factors for adherence long-term to exercise among non-ambulatory children with CP, ambulatory children with CP and non-disabled children, and furthermore a description of factors facilitating and hindering health and well-being.

ELIGIBILITY:
Inclusion Criteria:

* non-ambulatory children with CP defined as GMFCS-E&R IV-V, ambulatory children with CP defined as GMFCS-E&R I-II and healthy controls: non-disabled children not participating in any regular and planned physical exercise.

Exclusion Criteria:

* Ambulatory children with CP walking with a walking aid (GMFCS-E&R III); non-disabled children with other neurological diagnoses, metabolic diagnoses, orthopaedic disabilities, asthma, heart diseases, cognitive impairments or indigestion of regular medication.

Ages: 10 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2019-05-01 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Brain derived neurotropic factor (BDNF) | 12 months

SECONDARY OUTCOMES:
Nerve growth factor (NGF) | 12 months
Vascular endothelial growth factor (VEGF) | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Health Sciences Centre, Lund, Skåne County, Sweden

IPD SHARING:
Plan to Share IPD: No